CLINICAL TRIAL: NCT07301333
Title: A Phase 1 Study To Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and the Effect of Food on the Bioavailability of HRS-6257 in Healthy Subjects
Brief Title: A Study of Single and Multiple Doses of HRS-6257 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-6257-101
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-6257 group (Experimental)
  Interventions: Drug: HRS-6257
- placebo group (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HRS-6257 — HRS-6257
  Arms: HRS-6257 group
Drug: placebo — placebo
  Arms: placebo group

SUMMARY:
This is a phase I, randomised, single-blind placebo-controlled, 2-part study to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and food effect of single and multiple oral doses of HRS-6257 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 55 years old (based on the time of signing the informed consent form), both males and females are eligible.
2. The body weight of males ≥ 50 kg, and that of females ≥ 45 kg, and body mass index (BMI): 19 - 28 kg/m².
3. Female subjects must be non-pregnant or non-childbearing potential;
4. Subjects must understand the study procedures and methods, voluntarily participate in this study and sign the ICF in person.

Exclusion Criteria:

1. History of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological disease;
2. Known or suspected hypersensitivity to trial product(s) or related products;
3. 12-lead ECG demonstrating QTcF >450 msec or history or risk factors for QT prolongation;
4. Blood donation of more than 200 mL within the last 6 months
5. Use of prescription or nonprescription drugs and dietary and herbal supplements within 14 days or 7 half-lives;
6. Positive screening tests for hepatitis B or C, HIV, alcohol, drugs of abuse.
7. Previous administration with an investigational product (drug or vaccine) within 3 months;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events | from ICF signing date to Day 14 or Day 21 or Day 27

SECONDARY OUTCOMES:
AUC of HRS-6257 | 0 hour to 72 hour after administration
Cmax of HRS-6257 | 0 hour to 72 hour after administration
Tmax of HRS-6257 | 0 hour to 72 hour after administration
t1/2 of HRS-6257 | 0 hour to 72 hour after administration
CL/F of HRS-6257 | 0 hour to 72 hour after administration
Vz/F of HRS-6257 | 0 hour to 72 hour after administration
Pain tolerance time for the Cold Pain Test | Day 1 to Day 1 or Day 14
Number of Participants With Clinically Meaningful Findings in Columbia Suicide Severity Rating Scale (C-SSRS) Responses | from ICF signing date to Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided